CLINICAL TRIAL: NCT04922892
Title: Total Parathyroidectomy With Autotransplantation Versus Total Parathyroidectomy Alone for Secondary Hyperparathyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOTAR-2021-05-31
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-05

CONDITIONS: Secondary Hyperparathyroidism;Parathyroidectomy
Keywords: Secondary Hyperparathyroidism;Parathyroidectomy;hemodialysis
MeSH Terms: interventions — Parathyroidectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Parathyroidectomy Alone (Experimental): Total Parathyroidectomy Alone , without autotransplantation
  Interventions: Procedure: Parathyroidectomy
- Total Parathyroidectomy With Autotransplantation (Active Comparator): Total Parathyroidectomy With Autotransplantation
  Interventions: Procedure: Parathyroidectomy

INTERVENTIONS:
Procedure: Parathyroidectomy — Total Parathyroidectomy With Autotransplantation or Total Parathyroidectomy Alone

SUMMARY:
Total parathyroidectomy with autotransplantation (TPTX+AT) and Total parathyr- oidectomy alone (TPTX) are the common surgical procedures.The purpose of the study was to compare the long-term benefits of surgery between the two groups.

DETAILED DESCRIPTION:
The trial was performed as a nonconfirmatory randomized controlled pilot trial with 200 patients on long-term dialysis with otherwise uncontrollable SHPT to generate data on the rate of recurrent disease within a 5-year follow-up period after TPTX or TPTX+AT. Parathyroid hormone (PTH) and calcium levels, recurrent or persistent hyperparathyroidism, parathyroid reoperations, morbidity, and mortality were evaluated during a 5-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

Severe renal secondary hyperparathyroidism

Exclusion Criteria:

Patients with diabetes a history of chronic inflammatory disease a history of malignant tumor a history of kidney transplantation a history of neck surgery a history of alcohol abuse a history of drug abuse inability to cooperate with the participants refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
the rate of recurrent | 60 months
  the rate of recurrent

CONTACTS AND LOCATIONS:
Overall Officials: Mingxia XIONG, Ph.D, Study Director — Nanjing Medcial university
Locations (1):
- NanjingMU, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schlosser K, Bartsch DK, Diener MK, Seiler CM, Bruckner T, Nies C, Meyer M, Neudecker J, Goretzki PE, Glockzin G, Konopke R, Rothmund M. Total Parathyroidectomy With Routine Thymectomy and Autotransplantation Versus Total Parathyroidectomy Alone for Secondary Hyperparathyroidism: Results of a Nonconfirmatory Multicenter Prospective Randomized Controlled Pilot Trial. Ann Surg. 2016 Nov;264(5):745-753. doi: 10.1097/SLA.0000000000001875. PMID 27741007
- [Result] Schlosser K, Veit JA, Witte S, Fernandez ED, Victor N, Knaebel HP, Seiler CM, Rothmund M. Comparison of total parathyroidectomy without autotransplantation and without thymectomy versus total parathyroidectomy with autotransplantation and with thymectomy for secondary hyperparathyroidism: TOPAR PILOT-Trial. Trials. 2007 Sep 18;8:22. doi: 10.1186/1745-6215-8-22. PMID 17877805
- [Result] Abruzzo A, Gioviale MC, Damiano G, Palumbo VD, Buscemi S, Lo Monte G, Gulotta L, Buscemi G, Lo Monte AI. Reoperation for persistent or recurrent secondary hyperparathyroidism. Acta Biomed. 2017 Oct 23;88(3):325-328. doi: 10.23750/abm.v88i3.4722. PMID 29083339
- [Result] Coulston JE, Egan R, Willis E, Morgan JD. Total parathyroidectomy without autotransplantation for renal hyperparathyroidism. Br J Surg. 2010 Nov;97(11):1674-9. doi: 10.1002/bjs.7192. PMID 20641052